CLINICAL TRIAL: NCT01193920
Title: A Phase Ib/II Randomized, Observer-Blind, Controlled, Single Centre Study of a Trivalent Group B Streptococcus Vaccine in Healthy Non-Pregnant Women Leading Into a Dose-Ranging Study in Pregnant Women in South Africa
Brief Title: Safety and Immunogenicity of a Group B Streptococcus Vaccine in Non Pregnant and Pregnant Women 18-40 Years of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V98_08; MCC Reference n° 20100601 (Other: South African authorities)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Streptococcal Infections
Keywords: Group B streptococcus; GBS; Vaccine; Prevention of group B streptococcus infection
MeSH Terms: conditions — Streptococcal Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- 1: GBS Trivalent Vaccine with aluminium - 20/20/20 μg (Experimental): Non-pregnant women who received two injections of 20/20/20 μg dose of Group B Streptococcus (GBS) Trivalent Vaccine with aluminum.
  Interventions: Biological: Group B Streptococcus Trivalent Vaccine - 20/20/20 μg
- 2: Placebo - Sterile saline (Placebo Comparator): Non-Pregnant Women who received two injection of saline solution.
  Interventions: Other: Saline solution
- 3: GBS Trivalent Vaccine - 0.5/0.5/0.5 µg (Experimental): Pregnant women who received one injection of 0.5/0.5/0.5 μg dose of non adjuvanted Group B Streptococcus (GBS) Trivalent Vaccine.
  Interventions: Biological: Group B Streptococcus Trivalent Vaccine - 0.5/0.5/0.5 μg
- 4: GBS Trivalent Vaccine - 2.5/2.5/2.5 µg (Experimental): Pregnant Women who received one injection of 2.5/2.5/2.5 μg dose of non adjuvanted Group B Streptococcus (GBS) Trivalent Vaccine.
  Interventions: Biological: Group B Streptococcus Trivalent Vaccine - 2.5/2.5/2.5 μg
- 5: GBS Trivalent Vaccine - 5/5/5 µg (Experimental): Pregnant women who received one injection of 5/5/5 μg dose of non adjuvanted Group B Streptococcus (GBS) Trivalent Vaccine.
  Interventions: Biological: Group B Streptococcus Trivalent Vaccine - 5/5/5 μg
- 6: Placebo - Sterile saline (Placebo Comparator): Pregnant Women who received one injection of saline solution.
  Interventions: Other: saline solution

INTERVENTIONS:
Biological: Group B Streptococcus Trivalent Vaccine - 20/20/20 μg — Subjects received two injections of 20/20/20 μg dose of Group B Streptococcus (GBS) Trivalent Vaccine with aluminum.
  Arms: 1: GBS Trivalent Vaccine with aluminium - 20/20/20 μg
Other: Saline solution — Subjects received two injection of saline solution.
  Arms: 2: Placebo - Sterile saline
Biological: Group B Streptococcus Trivalent Vaccine - 0.5/0.5/0.5 μg — Subjects received one injection of 0.5/0.5/0.5 μg dose of non adjuvanted Group B Streptococcus (GBS) Trivalent Vaccine.
  Arms: 3: GBS Trivalent Vaccine - 0.5/0.5/0.5 µg
Biological: Group B Streptococcus Trivalent Vaccine - 2.5/2.5/2.5 μg — Subjects received one injection of 2.5/2.5/2.5 μg dose of non adjuvanted Group B Streptococcus (GBS) Trivalent Vaccine.
  Arms: 4: GBS Trivalent Vaccine - 2.5/2.5/2.5 µg
Biological: Group B Streptococcus Trivalent Vaccine - 5/5/5 μg — Subjects received one injection of 5/5/5 μg dose of non adjuvanted Group B Streptococcus (GBS) Trivalent Vaccine.
  Arms: 5: GBS Trivalent Vaccine - 5/5/5 µg
Other: saline solution — Subjects received one injection of saline solution.
  Arms: 6: Placebo - Sterile saline

SUMMARY:
This study will evaluate the safety and immunogenicity of a Group B Streptococcus vaccine at one dose in healthy non pregnant women and then in three different doses in healthy pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (Non Pregnant Women): Healthy females 18-40 years of age inclusive.
* Group 2 (Healthy Pregnant Women): Healthy pregnant women 18-40 yrs of age (between 28-35 weeks gestation)

Exclusion Criteria:

* Group 1 (Non Pregnant Women): Pregnant or nursing; History of severe allergy to previous vaccines; Known HIV positive
* Group 2 (Healthy Pregnant Women): History of severe allergy to previous vaccines; Known HIV positive

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis
Locations (1):
- Chris Hani Baragwanath Hospital, Chris Hani Rd, Soweto, Johannesburg, South Africa

REFERENCES:
- [Derived] Madhi SA, Koen A, Cutland CL, Jose L, Govender N, Wittke F, Olugbosi M, Sobanjo-Ter Meulen A, Baker S, Dull PM, Narasimhan V, Slobod K. Antibody Kinetics and Response to Routine Vaccinations in Infants Born to Women Who Received an Investigational Trivalent Group B Streptococcus Polysaccharide CRM197-Conjugate Vaccine During Pregnancy. Clin Infect Dis. 2017 Nov 13;65(11):1897-1904. doi: 10.1093/cid/cix666. PMID 29029127
- [Derived] Madhi SA, Cutland CL, Jose L, Koen A, Govender N, Wittke F, Olugbosi M, Meulen AS, Baker S, Dull PM, Narasimhan V, Slobod K. Safety and immunogenicity of an investigational maternal trivalent group B streptococcus vaccine in healthy women and their infants: a randomised phase 1b/2 trial. Lancet Infect Dis. 2016 Aug;16(8):923-34. doi: 10.1016/S1473-3099(16)00152-3. Epub 2016 Apr 29. PMID 27139805
- [Derived] Cutland CL, Cunnington M, Olugbosi M, Jones SA, Hugo A, Maharaj K, Slobod K, Madhi SA. Lessons learnt from enrolment and follow up of pregnant women and their infants in clinical trials in South Africa, a low-middle income country. Vaccine. 2015 Nov 25;33(47):6406-12. doi: 10.1016/j.vaccine.2015.08.040. Epub 2015 Sep 26. PMID 26409812

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-pregnant 20/20/20 μg +Aluminum Hydroxide: Non-pregnant women who received two injections of 20/20/20 μg dose of trivalent GBS vaccine with aluminum
- Non-pregnant/Placebo: Non-pregnant women received two injections of saline solution
- Pregnant 0.5/0.5/0.5 μg: Pregnant women who received one injection of 0.5/0.5/0.5 μg dose of non adjuvanted trivalent GBS vaccine
- Pregnant 2.5/2.5/2.5 μg: Pregnant women who received one injection of 2.5/2.5/2.5 μg dose of non adjuvanted trivalent GBS vaccine
- Pregnant 5/5/5 μg: Pregnant women who received one injection of 5/5/5 μg dose of non adjuvanted trivalent GBS vaccine
- Pregnant/Placebo: Pregnant women who received one injection of saline solution
- Infants 0.5/0.5/0.5 μg: Infants born from women who received one injection of 0.5/0.5/0.5 μg dose of non adjuvanted trivalent GBS vaccine
- Infants 2.5/2.5/2.5 μg: Infants born from women who received one injection of 2.5/2.5/2.5 μg dose of non adjuvanted trivalent GBS vaccine
- Infants 5/5/5 μg: Infants born from women who received one injection of 5/5/5 μg dose of non adjuvanted trivalent GBS vaccine
- Infants / Placebo: Infants born from women who received saline solution
Period: Overall Study
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo | Infants 0.5/0.5/0.5 μg | Infants 2.5/2.5/2.5 μg | Infants 5/5/5 μg | Infants / Placebo
Started | 40 | 20 | 80 | 80 | 80 | 80 | 80 | 80 | 76 | 81
Completed | 37 | 20 | 74 | 76 | 74 | 76 | 74 | 76 | 71 | 74
Not Completed | 3 | 0 | 6 | 4 | 6 | 4 | 6 | 4 | 5 | 7
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 1 | 3 | 1 | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 3 | 3 | 1 | 0 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 4
Not completed — Unable to classify | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done on the all enrolled population.
Groups:
- Infants / Placebo: Infants born from women who received one injection of saline solution
- Total: Total of all reporting groups
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo | Infants 0.5/0.5/0.5 μg | Infants 2.5/2.5/2.5 μg | Infants 5/5/5 μg | Infants / Placebo | Total
Number analyzed (Participants) | 40 | 20 | 80 | 80 | 80 | 80 | 80 | 80 | 76 | 81 | 697
Age, Customized [Mean (Standard Deviation); unit: years]
  Non pregnant subjects | 28.6 (5.0) | 29.4 (5.1) | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | 28.8 (5.0)
  Maternal subjects | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | 25.3 (5.2) | 25.3 (5.2) | 24.2 (4.7) | 25.7 (5.4) | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | 25.1 (5.1)
Age, Customized [Mean (Standard Deviation); unit: days] | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | 3.0 (3.3) | 4.0 (7.8) | 5.5 (16.9) | 3.5 (8.8) | 4.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 80 | 80 | 80 | 80 | 45 | 38 | 33 | 48 | 544
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 42 | 43 | 33 | 153
Region of Enrollment [Number; unit: participants]
  South Africa | 40 | 20 | 80 | 80 | 80 | 80 | 80 | 80 | 76 | 81 | 697

OUTCOME MEASURES:

1. Primary Outcome: The Percentages of Non-pregnant Subjects With Antibody Concentrations Above a Defined Threshold at One Month After the Second Vaccination.
Description: The percentages of non-pregnant subjects with antibody concentrations above a defined threshold per serotype after the administration of two vaccine doses administered one month apart. Defined thresholds for antibody concentrations, which exceed pre-defined serotype specific ELISA values are 1, 2, 3, 5 and 8 μg/mL.
Time Frame: Day 61, one month after the second vaccination
Population: Full Analysis Set (FAS) - primary, non-pregnant subjects, i.e. all enrolled subjects who provided at least one evaluable serum sample result at Day 1 (prior to vaccination) and Day 61
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo
Number analyzed (Participants) | 35 | 19
percentage of subjects
  Serotype Ia >=1 μg/mL (N=34, 19) | 91 [76 to 98] | 37 [16 to 62]
  Serotype Ia >=2 μg/mL (N=34, 19) | 91 [76 to 98] | 32 [13 to 57]
  Serotype Ia >=3 μg/mL (N=34, 19) | 88 [73 to 97] | 26 [9 to 51]
  Serotype Ia >=5 μg/mL (N=34, 19) | 79 [62 to 91] | 16 [3 to 40]
  Serotype Ia >=8 μg/mL (N=34, 19) | 76 [59 to 89] | 16 [3 to 40]
  Serotype Ib >=1 μg/mL (N=33, 17) | 73 [54 to 87] | 24 [7 to 50]
  Serotype Ib >=2 μg/mL (N=33, 17) | 67 [48 to 82] | 12 [1 to 36]
  Serotype Ib >=3 μg/mL (N=33, 17) | 64 [45 to 80] | 6 [0 to 29]
  Serotype Ib >=5 μg/mL (N=33, 17) | 42 [25 to 61] | 6 [0 to 29]
  Serotype Ib >=8 μg/mL (N=33, 17) | 39 [23 to 58] | 6 [0 to 29]
  Serotype III >=1 μg/mL | 89 [73 to 97] | 37 [16 to 62]
  Serotype III >=2 μg/mL | 69 [51 to 83] | 21 [6 to 46]
  Serotype III >=3 μg/mL | 63 [45 to 79] | 21 [6 to 46]
  Serotype III >=5 μg/mL | 51 [34 to 69] | 11 [1 to 33]
  Serotype III >=8 μg/mL | 49 [31 to 66] | 5 [0 to 26]

2. Primary Outcome: Antibody Geometric Mean Concentrations (GMC) in Non-pregnant Women at One Month After the Second Vaccination.
Description: Antibody GMC per serotype in non-pregnant women after receiving two doses of the study vaccine administered one month apart .
Time Frame: Day 61, one month after the second vaccination
Population: FAS - primary, non-pregnant subjects
Measure: Geometric Mean (95% Confidence Interval); unit: concentrations (μg/mL)
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo
Number analyzed (Participants) | 35 | 19
concentrations (μg/mL)
  Serotype Ia (N=34, 19) | 40 [26 to 62] | 0.88 [0.49 to 1.59]
  Serotype Ib (N=33, 17) | 5.3 [2.94 to 9.56] | 0.25 [0.12 to 0.55]
  Serotype III | 11 [6.43 to 19] | 0.61 [0.29 to 1.27]

3. Secondary Outcome: The Percentages of Maternal Subjects With Antibody Concentrations Above a Defined Threshold Per Serotype at One Month After Vaccination.
Description: The percentages of maternal subjects with antibody concentrations above a defined threshold per serotype at one month after the administration of one of three different doses of the study vaccine or placebo. Antibody concentrations which exceed pre-defined serotype specific ELISA values are 1, 2, 3, 5 and 8 μg/mL.
Time Frame: Day 31, one month after vaccination
Population: FAS, secondary, maternal subjects, day 31, i.e. all enrolled subjects who provided at least one evaluable serum sample result at day 1 (prior to vaccination) and at day 31
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo
Number analyzed (Participants) | 75 | 74 | 69 | 76
percentage of subjects
  serotype Ia>=1μg/mL (N=75, 74, 69, 75) | 85 [75 to 92] | 77 [66 to 86] | 88 [78 to 95] | 33 [23 to 45]
  serotype Ia>=2μg/mL (N=75, 74, 69, 75) | 79 [68 to 87] | 77 [66 to 86] | 81 [70 to 90] | 27 [17 to 38]
  serotype Ia>=3μg/mL (N=75, 74, 69, 75) | 76 [65 to 85] | 73 [61 to 83] | 78 [67 to 87] | 23 [14 to 34]
  serotype Ia>=5μg/mL (N=75, 74, 69, 75) | 75 [63 to 84] | 70 [59 to 80] | 71 [59 to 81] | 15 [8 to 25]
  serotype Ia>=8μg/mL (N=75, 74, 69, 75) | 71 [59 to 81] | 70 [59 to 80] | 71 [59 to 81] | 9 [4 to 18]
  serotype Ib>=1μg/mL (N= 65, 69, 66, 61) | 65 [52 to 76] | 68 [56 to 79] | 62 [49 to 74] | 21 [12 to 34]
  serotype Ib>=2μg/mL (N= 65, 69, 66, 61) | 60 [47 to 72] | 54 [41 to 66] | 50 [37 to 63] | 13 [6 to 24]
  serotype Ib>=3μg/mL (N= 65, 69, 66, 61) | 54 [41 to 66] | 48 [36 to 60] | 44 [32 to 57] | 11 [5 to 22]
  serotype Ib>=5μg/mL (N= 65, 69, 66, 61) | 48 [35 to 60] | 43 [32 to 56] | 36 [25 to 49] | 10 [4 to 20]
  serotype Ib>=8μg/mL (N= 65, 69, 66, 61) | 43 [31 to 56] | 39 [28 to 52] | 30 [20 to 43] | 8 [3 to 18]
  serotype III>=1μg/mL (N= 73, 74, 68, 76) | 70 [58 to 80] | 65 [53 to 76] | 57 [45 to 69] | 13 [6 to 23]
  serotype III>=2μg/mL (N=73, 74, 68, 76) | 58 [45 to 69] | 54 [42 to 66] | 51 [39 to 64] | 12 [6 to 21]
  serotype III>=3μg/mL (N=73, 74, 68, 76) | 48 [36 to 60] | 50 [38 to 62] | 44 [32 to 57] | 4 [1 to 11]
  serotype III>=5μg/mL (N=73, 74, 68, 76) | 41 [30 to 53] | 43 [32 to 55] | 32 [22 to 45] | 3 [0 to 9]
  serotype III>=8μg/mL (N=73, 74, 68, 76) | 38 [27 to 50] | 34 [23 to 46] | 29 [19 to 42] | 3 [0 to 9]

4. Primary Outcome: The Percentages of Maternal Subjects With Antibody Concentrations Above a Defined Threshold at Day of Delivery.
Description: The percentages of maternal subjects with antibody concentrations above a defined threshold per serotype following the administration of one of three different doses of the study vaccine or placebo.Antibody concentrations which exceed pre-defined serotype specific ELISA values are 1, 2, 3, 5 and 8 μg/mL.
Time Frame: Day of delivery
Population: FAS primary, maternal subjects, i.e. all enrolled subjects who provided at least one evaluable serum sample result at day 1 (prior to vaccination) and at delivery
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo
Number analyzed (Participants) | 76 | 77 | 73 | 78
percentage of subjects
  Serotype Ia >= 1 μg/mL (N=76,77, 73, 76) | 86 [76 to 93] | 83 [73 to 91] | 89 [80 to 95] | 38 [27 to 50]
  Serotype Ia >= 2 μg/mL (N=76, 77, 73, 76) | 78 [67 to 86] | 74 [63 to 83] | 81 [70 to 89] | 26 [17 to 38]
  Serotype Ia >= 3 μg/mL (N=76, 77, 73, 76) | 75 [64 to 84] | 71 [60 to 81] | 77 [65 to 86] | 21 [13 to 32]
  Serotype Ia >= 5 μg/mL (N=76, 77, 73, 76) | 72 [61 to 82] | 69 [57 to 79] | 75 [64 to 85] | 18 [10 to 29]
  Serotype Ia >= 8 μg/mL (N=76, 77, 73, 76) | 64 [53 to 75] | 64 [52 to 74] | 71 [59 to 81] | 9 [4 to 18]
  Serotype Ib >= 1 μg/mL (N=69, 74, 71, 58) | 58 [45 to 70] | 65 [53 to 76] | 65 [53 to 76] | 14 [6 to 25]
  Serotype Ib >= 2 μg/mL (69, 74, 71, 58) | 52 [40 to 64] | 51 [39 to 63] | 48 [36 to 60] | 10 [4 to 21]
  Serotype Ib >= 3 μg/mL (N=69, 74, 71, 58) | 43 [32 to 56] | 49 [37 to 61] | 42 [31 to 55] | 10 [4 to 21]
  Serotype Ib >= 5 μg/mL (N=69, 74, 71, 58) | 41 [29 to 53] | 41 [29 to 53] | 37 [25 to 49] | 9 [3 to 19]
  Serotype Ib >= 8 μg/mL (N=69, 74, 71, 58) | 36 [25 to 49] | 36 [26 to 48] | 32 [22 to 45] | 3 [0 to 12]
  Serotype Ill >= 1 μg/mL (N=74, 77, 73, 78) | 69 [57 to 79] | 66 [55 to 77] | 64 [52 to 75] | 14 [7 to 24]
  Serotype Ill >= 2 μg/mL (N=74, 77, 73, 78) | 62 [50 to 73] | 53 [42 to 65] | 51 [39 to 63] | 9 [4 to 18]
  Serotype Ill >= 3 μg/mL (N=74, 77, 73, 78) | 49 [37 to 61] | 44 [33 to 56] | 42 [31 to 55] | 4 [1 to 11]
  Serotype Ill >= 5 μg/mL (N=74, 77, 73, 78) | 39 [28 to 51] | 49 [29 to 52] | 36 [25 to 48] | 3 [0 to 9]
  Serotype Ill >= 8 μg/mL (N=74, 77, 73, 78) | 34 [23 to 46] | 35 [25 to 47] | 29 [19 to 41] | 3 [0 to 9]

5. Primary Outcome: Antibody GMC in Maternal Subjects at Day of Delivery
Description: Antibody GMC per serotype in maternal subjects at day of delivery following one administration of one of three different doses of the study vaccine or placebo are reported.
Time Frame: Day of delivery
Population: FAS primary, maternal subjects
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration (μg/mL)
Arm/Group | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo
Number analyzed (Participants) | 76 | 77 | 73 | 78
Concentration (μg/mL)
  Serotype Ia (N= 76, 77, 73, 76) | 9.95 [6.6 to 15] | 14 [9.19 to 21] | 24 [16 to 36] | 0.67 [0.46 to 0.99]
  Serotype Ib (N=69, 74, 71, 58) | 2.5 [1.61 to 3.88] | 4.3 [2.74 to 6.76] | 2.93 [1.79 to 4.77] | 0.38 [0.25 to 0.59]
  Serotype III (N=74, 77, 73, 78) | 2.63 [1.8 to 3.85] | 3.66 [2.52 to 5.31] | 2.83 [1.92 to 4.17] | 0.25 [0.18 to 0.34]

6. Secondary Outcome: Antibody GMC Per Serotype in Maternal Subjects at One Month After Vaccination
Description: Antibody GMC per serotype in maternal subjects at one month after the administration of one of three different doses of the study vaccine or placebo.
Time Frame: day 31
Population: FAS, secondary, maternal subjects, day 31
Measure: Geometric Mean (95% Confidence Interval); unit: concentration (μg/mL)
Arm/Group | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo
Number analyzed (Participants) | 75 | 74 | 69 | 76
concentration (μg/mL)
  serotype Ia (N=75, 74, 69, 75) | 13 [8.27 to 21] | 15 [9.54 to 25] | 26 [16 to 43] | 0.62 [0.41 to 0.93]
  serotype Ib (N=65, 69, 66, 61) | 2.78 [1.68 to 4.59] | 5.42 [3.21 to 9.18] | 3.66 [2.06 to 6.52] | 0.3 [0.19 to 0.49]
  serotype III (N=73, 74, 68, 76) | 3.01 [1.96 to 4.62] | 4.11 [2.68 to 6.31] | 2.77 [1.75 to 4.37] | 0.19 [0.13 to 0.27]

7. Secondary Outcome: The Percentage of Non-pregnant Subjects With Antibody Concentrations Above a Defined Threshold at One Year After the First Vaccination.
Description: The percentage of non-pregnant subjects with antibody concentrations above a defined threshold per serotype after the administration of two vaccine doses one month apart. Antibody concentrations which exceed pre-defined serotype specific ELISA values are 1, 2, 3, 5 and 8 mcg/mL.
Time Frame: Day 361, one year after the first vaccination
Population: FAS persistence, non-pregnant subjects, i.e. all enrolled subjects who provided at least one evaluable serum sample result at day 1 (prior to vaccination) and day 361.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo
Number analyzed (Participants) | 37 | 20
percentage of subjects
  Serotype Ia >=1μg/mL | 86 [71 to 95] | 30 [12 to 54]
  Serotype Ia >=2μg/mL | 76 [59 to 88] | 30 [12 to 54]
  Serotype Ia >=3μg/mL | 76 [59 to 88] | 25 [9 to 49]
  Serotype Ia >=5μg/mL | 70 [53 to 84] | 15 [3 to 38]
  Serotype Ia >=8μg/mL | 62 [45 to 78] | 10 [1 to 32]
  Serotype Ib >=1μg/mL (N=37, 19) | 81 [65 to 92] | 21 [6 to 46]
  Serotype Ib >=2μg/mL (N=37, 19) | 65 [47 to 80] | 16 [3 to 40]
  Serotype Ib >=3μg/mL (37, 19) | 62 [45 to 78] | 5 [0 to 26]
  Serotype Ib >=5μg/mL (N=37, 19) | 38 [22 to 55] | 5 [0 to 26]
  Serotype Ib >=8μg/mL (N=37, 19) | 32 [18 to 50] | 5 [0 to 26]
  Serotype III >=1μg/mL | 81 [65 to 92] | 20 [6 to 44]
  Serotype III >=2μg/mL | 70 [53 to 84] | 15 [3 to 38]
  Serotype III >=3μg/mL | 65 [47 to 80] | 15 [3 to 38]
  Serotype III >=5μg/mL | 54 [37 to 71] | 5 [0 to 25]
  Serotype III >=8μg/mL | 41 [25 to 58] | 5 [0 to 25]

8. Secondary Outcome: Antibody GMC in Non-pregnant Subjects at One Year After the First Vaccination
Description: Antibody GMC per serotype in non-pregnant subjects after receiving two doses of the study vaccine administered one month apart, at one year after first vaccination.
Time Frame: Day 361, one year after the first vaccination
Population: FAS persistence, non-pregnant subjects
Measure: Geometric Mean (95% Confidence Interval); unit: concentration (μg/mL)
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo
Number analyzed (Participants) | 37 | 20
concentration (μg/mL)
  serotype Ia | 15 [9.86 to 22] | 0.86 [0.51 to 1.45]
  serotype Ib (N=37, 19) | 5.28 [3.49 to 7.98] | 0.4 [0.23 to 0.69]
  serotype III | 7.03 [4.5 to 11] | 0.3 [0.17 to 0.55]

9. Secondary Outcome: Number of Non-pregnant Subjects Reporting Solicited and Unsolicited Adverse Events
Description: Number of non-pregnant subjects reporting solicited and unsolicited adverse events following 2 injections (1 month apart) of the trivalent GBS vaccine at a dose of 20/20/20 μg with aluminum at one month after second vaccination are reported.
Time Frame: Day 61
Population: Safety set, solicited and unsolicited reactogenicity, non-pregnant subjects
Measure: Number; unit: participants
Groups:
- Non Pregnant/Placebo: Non pregnant women received two injections of saline solution
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non Pregnant/Placebo
Number analyzed (Participants) | 40 | 20
participants
  Solicited adverse events | 40 | 19
  Unsolicited adverse events | 30 | 16

10. Secondary Outcome: Number of Maternal Subjects Reporting Solicited and Unsolicited Adverse Events
Description: Number of maternal subjects reporting solicited and unsolicited adverse events following the administration of either one of three different doses of the study vaccine or placebo.
Time Frame: From day 1 to one year after delivery
Population: Safety set, solicited and unsolicited reactogenicity, maternal subjects
Measure: Number; unit: participants
Arm/Group | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo
Number analyzed (Participants) | 80 | 80 | 80 | 80
participants
  solicited adverse events (N=80, 80, 79, 80) | 59 | 46 | 59 | 57
  unsolicited adverse events | 70 | 59 | 62 | 69

11. Secondary Outcome: Antibody GMC Per Serotype at Different Time Points in Infants
Description: Antibody GMC per serotype on the day of birth, at 6 weeks and 3 months of age in infants born from women who received either one of three different doses of the study vaccine or placebo.
Time Frame: Day 4, day 43 and day 91 after birth
Population: Per Protocol Set, infants, i.e. all subjects who provided evaluable serum samples at birth, study day 43, study day 91 and within the required time frames
Measure: Geometric Mean (95% Confidence Interval); unit: concentration (μg/mL)
Arm/Group | Infants 0.5/0.5/0.5 μg | Infants 2.5/2.5/2.5 μg | Infants 5/5/5 μg | Infants / Placebo
Number analyzed (Participants) | 75 | 77 | 69 | 76
concentration (μg/mL)
  Serotype Ia (day 4; N=75, 76, 69, 73) | 6.66 [4.03 to 11] | 6.52 [3.96 to 11] | 12 [7.21 to 20] | 0.49 [0.34 to 0.71]
  Serotype Ia (day 43; N= 75, 76, 68, 71) | 3.21 [2.01 to 5.13] | 2.95 [1.85 to 4.7] | 5.54 [3.38 to 9.06] | 0.31 [0.23 to 0.42]
  Serotype Ia (day 91; N=71, 75, 64, 75) | 1.97 [1.31 to 2.95] | 2.22 [1.49 to 3.29] | 2.78 [1.81 to 4.26] | 0.38 [0.29 to 0.49]
  Serotype Ib (day 4; N=71, 71, 66, 62) | 1.15 [0.68 to 1.95] | 1.72 [1.02 to 2.92] | 1.39 [0.81 to 2.4] | 0.21 [0.14 to 0.32]
  Serotype Ib (day 43; N=72, 77, 67, 69) | 0.73 [0.47 to 1.14] | 0.88 [0.57 to 1.35] | 0.67 [0.42 to 1.07] | 0.15 [0.11 to 0.21]
  Serotype Ib (day 91; N= 74, 73, 66, 76) | 0.85 [0.61 to 1.18] | 1.08 [0.77 to 1.51] | 0.83 [0.59 to 1.19] | 0.5 [0.39 to 0.63]
  Serotype III (day 4; N= 57, 64, 58, 52) | 2.11 [1.26 to 3.54] | 2.3 [1.41 to 3.76] | 1.72 [1.03 to 2.87] | 0.29 [0.19 to 0.43]
  Serotype III (day 43; N= 64, 75, 61, 63) | 0.82 [0.53 to 1.27] | 0.88 [0.59 to 1.31] | 0.68 [0.43 to 1.06] | 0.16 [0.12 to 0.22]
  Serotype III (day 91; N= 63, 63, 57, 69) | 0.6 [0.42 to 0.85] | 0.69 [0.48 to 0.98] | 0.51 [0.35 to 0.74] | 0.27 [0.21 to 0.34]

12. Secondary Outcome: Number of Infants Reporting Serious Adverse Events
Description: Number of infants born from women who received either one of three different doses of the study vaccine or placebo who reported serious adverse events
Time Frame: one year after birth
Measure: Number; unit: Number of subjects
Arm/Group | Infants 0.5/0.5/0.5 μg | Infants 2.5/2.5/2.5 μg | Infants 5/5/5 μg | Infants / Placebo
Number analyzed (Participants) | 79 | 79 | 74 | 78
Number of subjects
  Serious AEs | 19 | 13 | 13 | 18
  At least possibly related SAEs | 0 | 0 | 0 | 0
  AEs leading to withdrawal | 1 | 2 | 0 | 1
  AEs leading to death | 1 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from day 1 to 7 after vaccination; unsolicited AEs and SAEs were collected from day 1 to day 361.
Description: Analyses was done on the Safety Population. Solicited AEs were collected through systematic assessment, unsolicited AEs were collected through non-systematic assesment.
Arm/Group | Non-pregnant 20/20/20 μg +Aluminum Hydroxide | Non-pregnant/Placebo | Pregnant 0.5/0.5/0.5 μg | Pregnant 2.5/2.5/2.5 μg | Pregnant 5/5/5 μg | Pregnant/Placebo | Infants 0.5/0.5/0.5 μg | Infants 2.5/2.5/2.5 μg | Infants 5/5/5 μg | Infants / Placebo
Serious Adverse Events (participants affected / at risk) | 2/40 | 1/20 | 27/80 | 24/80 | 25/80 | 30/80 | 19/79 | 13/79 | 13/74 | 18/78
Other Adverse Events (participants affected / at risk) | 40/40 | 19/20 | 72/80 | 67/80 | 70/80 | 71/80 | 44/79 | 49/79 | 48/74 | 51/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-pregnant 20/20/20 μg +Aluminum Hydroxide (N=40) | Non-pregnant/Placebo (N=20) | Pregnant 0.5/0.5/0.5 μg (N=80) | Pregnant 2.5/2.5/2.5 μg (N=80) | Pregnant 5/5/5 μg (N=80) | Pregnant/Placebo (N=80) | Infants 0.5/0.5/0.5 μg (N=79) | Infants 2.5/2.5/2.5 μg (N=79) | Infants 5/5/5 μg (N=74) | Infants / Placebo (N=78)
anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia foetal (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
congenital pneumonia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
strabism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 3
bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
bullous impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
chorioamnionitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
eczema herpeticum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 3 | 3
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
postpartum sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 1
streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
umbilical sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 0
urinary tract infection bacteria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
wound sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
perineal laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
coagulation factor IX level decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
convulsion neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 3
low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 2 | 1 | 5 | 0 | 0 | 0 | 0
eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 4 | 4 | 0 | 0 | 0 | 0 | 0
false labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 10 | 4 | 9 | 11 | 0 | 0 | 0 | 0
foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 4 | 2 | 12 | 0 | 0 | 0 | 0
haemorrage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
labour complication (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
postpartum haemorrage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 0 | 0 | 0
pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0
premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0
premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 6 | 4 | 1 | 5 | 0 | 0 | 0 | 0
prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
retained product of conception (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
vaginal haemorrage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
neonathal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 4
erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
labour induction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
subgaleal haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-pregnant 20/20/20 μg +Aluminum Hydroxide (N=40) | Non-pregnant/Placebo (N=20) | Pregnant 0.5/0.5/0.5 μg (N=80) | Pregnant 2.5/2.5/2.5 μg (N=80) | Pregnant 5/5/5 μg (N=80) | Pregnant/Placebo (N=80) | Infants 0.5/0.5/0.5 μg (N=79) | Infants 2.5/2.5/2.5 μg (N=79) | Infants 5/5/5 μg (N=74) | Infants / Placebo (N=78)
anaemia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 17 | 6 | 16 | 7 | 17 | 8 | 0 | 0 | 0 | 0
chills (General disorders) | 15 | 6 | 16 | 7 | 8 | 9 | 0 | 0 | 0 | 0
fatigue (General disorders) | 29 | 12 | 39 | 34 | 43 | 37 | 0 | 0 | 0 | 0
feeling hot (General disorders) | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
injection site induration (General disorders) | 19 | 4 | 7 | 9 | 9 | 3 | 0 | 0 | 0 | 0
injection site erythema (General disorders) | 12 | 3 | 10 | 8 | 7 | 2 | 0 | 0 | 0 | 0
injection site haemorrhage (General disorders) | 7 | 3 | 1 | 4 | 3 | 2 | 0 | 0 | 0 | 0
injection site pain (General disorders) | 39 | 15 | 28 | 25 | 26 | 24 | 0 | 0 | 0 | 0
injection site swelling (General disorders) | 14 | 2 | 2 | 5 | 5 | 1 | 0 | 0 | 0 | 0
injection site warmth (General disorders) | 24 | 9 | 21 | 12 | 15 | 15 | 0 | 0 | 0 | 0
malaise (General disorders) | 14 | 7 | 14 | 13 | 17 | 16 | 0 | 0 | 0 | 0
pain (General disorders) | 10 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
pyrexia (General disorders) | 6 | 0 | 5 | 1 | 4 | 2 | 0 | 0 | 0 | 0
influenza (Infections and infestations) | 1 | 1 | 8 | 2 | 15 | 5 | 0 | 1 | 1 | 0
tonsillitis (General disorders) | 3 | 0 | 0 | 4 | 4 | 3 | 0 | 0 | 0 | 0
upper respiratory tract infection (Infections and infestations) | 3 | 1 | 26 | 26 | 34 | 32 | 21 | 26 | 18 | 24
urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 4 | 7 | 8 | 0 | 0 | 0 | 1
aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 6 | 20 | 14 | 15 | 20 | 0 | 0 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 29 | 11 | 20 | 23 | 26 | 19 | 0 | 0 | 0 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 5 | 5 | 0 | 0 | 0 | 0
headache (Nervous system disorders) | 28 | 15 | 47 | 25 | 44 | 34 | 0 | 0 | 0 | 0
vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 2 | 6 | 9 | 7 | 0 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 3 | 7 | 6 | 1 | 1 | 1 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 4 | 6 | 9 | 17 | 20 | 15
rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 3 | 5 | 0 | 1 | 1 | 2 | 1
hypertension (Vascular disorders) | 3 | 0 | 4 | 3 | 6 | 6 | 0 | 0 | 0 | 0
induration (General disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 6 | 7 | 3
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 4 | 3 | 3
jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 5 | 2
bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 3
fungal skin infection (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 2 | 9 | 10 | 10 | 6
gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 2 | 1 | 1 | 6 | 7 | 1 | 3
oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 4
dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 11 | 6 | 4 | 6
dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 8 | 6
eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 5 | 12
Influenza like illness (General disorders) | 1 | 0 | 2 | 1 | 0 | 8 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement: the terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.